CLINICAL TRIAL: NCT05505877
Title: A Multicenter, Open-Label Phase 1/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics and Efficacy of BR790 Tablets in Combination With Tislelizumab Injection in Patients With Advanced Solid Tumors
Brief Title: Phase I/IIa Study of BR790 in Combination With Tislelizumab in Adult Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Gopherwood Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BR790-102
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumor
Keywords: BR790,SHP2, checkpoint inhibitor, PD-1, NSCLC, CRC, HNSCC
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR790+Tislelizumab dose escalation (Experimental): Dose escalation part
  Interventions: Drug: BR790+Tislelizumab
- BR790+Tislelizumab dose expansion (Experimental): Dose expansion part
  Interventions: Drug: BR790+Tislelizumab

INTERVENTIONS:
Drug: BR790+Tislelizumab — BR790 will be administered orally, variable dose.
  Tislelizumab will be administered as an intravenous infusion,fixed dose.

SUMMARY:
This study is a Phase I/IIa, multi-center, open-label study of BR790 in combination with Tislelizumab with a dose escalation part followed by a dose expansion part in adult subjects with advanced solid tumors.

These treatment to characterize the safety, tolerability, PK, PD and preliminary antitumor activity.

The study treatment will be administered until the subject experiences unacceptable toxicity, progressive disease, and/or has treatment discontinued at the discretion of the Investigator or the subject, or due to withdrawal of consent.

DETAILED DESCRIPTION:
Phase 1 (Dose Escalation Phase of BR790 Tablets Combined with Tislelizumab Injection): According to the incidence of DLT in BR790 Tablets Combined with Tislelizumab Injection Monoclonal Antibody in the Treatment of Advanced Solid Tumors, MTD and the Phase 2 clinical trial dose (RP2D) combining PK , efficacy and safety data were determined.

Stage II (BR790 Tablets combined with tislelizumab injection dose expansion stage): Evaluate the objective response rate (ORR) of BR790 Tablets combined with tislelizumab injection according to Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 .

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent voluntarily.
2. Age ≥18 and ≤75 years old.
3. Subjects with advanced solid tumors diagnosed by histology or cytology，whose desease progressed after standard treatment or have no standard treatment.
4. Had at least one measurable lesion.
5. ECOG≤1.
6. Expected survival period ≥ 3 months.

Exclusion Criteria:

1. Any previous treatment with SHP-2 inhibitor.
2. Symptomatic brain metastases.
3. Subjects with thoracic/ascites fluid that need drainage or intervention.
4. Subjects with not enough organ functional reserve at baseline, which met at least one of the following criteria： ANC<1.5×10^9/L PLT<100×10^9/L Hb<90g/L TBIL>1.5×ULN ALT, AST>2.5×ULN (without liver metastases) or ALT, AST>5×ULN (with liver metastases), Cr >1.5×ULN.
5. With uncontrolled severe disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 24 months
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle. (Dose escalation phase)
maximum tolerated dose (MTD) | 24 months
  Measurements of MTD (i.e. the highest dose of BR790 associated with the occurrence of Dose Limiting Toxicities (DLTs) in <33% of patients)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | 24 months
  Area under the plasma concentration time curve of BR790
Plasma concentration (Cmax) | 24 months
  Highest observed plasma concentration of BR790
t1/2 | 24 months
  Half life of BR790
Duration of response ( DCR ) | 24 months
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD). (Dose escalation phase)
Duration of response ( DOR ) | 24 months
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first. (Dose escalation phase)
Progression-free survival (PFS) | 24 months
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first. (Dose escalation phase)
Overall survival (OS) | 24 months
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor(Dose escalation phase)

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No